CLINICAL TRIAL: NCT06945081
Title: Wilson's Disease Treated With D-Penicillamine: Characterization of Skin Damage Secondary to Treatment by Measuring Skin Elasticity
Acronym: WILDERME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25CH057; ANSM (Other: 2025-A00509-40)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wilson Disease; D-Penicillamine; Effect of D-penicilline on Cutaneous Elastity of Wilson's Patient
Keywords: Cutaneous elastopathy
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: Exploratory, prospective, matched-control study. Cohort of Wilson's disease patients undergoing treatment with D-Penicillamine matched for age and sex to a control patient, as we know that skin elasticity is modified according to the patient's age and sex. This will enable us to study primarily the effect of treatment and its duration, although we know that other factors may come into play (sun exposure, smoking/alcohol consumption, etc.).
  Characterization of cutaneous side-effects of treatment by measuring skin tension lines (using a silicone mold on a small part of the skin of the forearm and cheek, enabling precise measurement of the tension lines, reproduced in these molds, by a confocal laser).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-penicillamine (Experimental): Patients with Wilson's disease treated with D-penicillamine for various exposure times
  Interventions: Other: Preparation of forearm molds with SILFLO® silicone
- Healthy patients (Active Comparator): Patients not diagnosed with wilson's disease and not receiving treatment that may affect skin elasticity
  Interventions: Other: Preparation of forearm molds with SILFLO® silicone

INTERVENTIONS:
Other: Preparation of forearm molds with SILFLO® silicone — Preparation of forearm molds with SILFLO® silicone (MONADERM, Monaco), CE-marked and already used routinely in dermocosmetics. These molds will, then, be analyzed.

SUMMARY:
Wilson's disease is a genetic disorder, resulting from an anomaly present on the ATP7B gene located on chromosome 13, causing a progressive accumulation of copper in various organs such as the liver, nervous system and cornea, leading to various hepatic and neurological disorders and a systemic evolution.

Currently, the first-line treatment for this disease is D-Penicillamine, which acts by chelation and promotes copper excretion through the urine. Unfortunately, this treatment also has significant side-effects, particularly on the skin. However, the pathogenesis of elastopathy in patients with Wilson's disease has yet to be fully characterized, and needs to be better understood in order to adapt the therapeutic strategy.

A silicon mold will be made on Wilson's disease patients, enabling the skin micro-relief to be shaped, and analyzed by confocal laser in comparison with the skin of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Diseased patients :

* Patient over 12 years old
* Patient with Wilson's disease confirmed by genetic analysis
* Patient followed up in the Wilson's Disease Reference Center for his care
* Patient treated with D-Penicillamine
* Patient with no other known elastic tissue pathology

Healthy volunteers :

* Patient over 12 years old
* Patient followed up in the dermatology department of St Etienne University Hospital
* Patient matched on sex and age with a patient from the "Wilson's disease" group
* Patient with no elastic tissue pathology

All patients :

* Patient affiliated to a national social security
* Patient with written informed consent

Exclusion Criteria:

All patients:

* Patient not taking a treatment (at investigator's discretion) that may modify skin elasticity
* Patient with pathological lesion(s) on forearm or cheek
* Patient with a potentially active/rejuvenative forearm or cheek treatment
* Patient having applied cream and/or make-up to the areas to be molded (forearm and cheek)
* Patient under guardianship
* Patient unable to follow study procedures
* Pregnant or breast-feeding women

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Skin tension measurement | At inclusion
  Measurement of skin tension indices on a silicone cast of the inner forearm with a confocal laser expressed as a percentage (from 0 (perfect tension balance) to 100 (absolute imbalance on one tension axis)) of patients treated with D-Penicillamine and healthy patients.

SECONDARY OUTCOMES:
Skin tension indices measurement on silicone casts | Year 1
  Measurement of skin tension indices on silicone casts of the inner and outer forearm with confocal laser and comparison between different groups of patients according to duration of exposure to treatment in subgroups: (< to 5 years, 5 to 10 years, 10 to 15 years and 15 years and more).
Skin tension indice measurement with confocal laser | Year 1
  Measurement of skin tension indices on various silicone casts of the inner and outer forearm and cheek with confocal laser and comparison between patients and age- and sex-matched control group patients

CONTACTS AND LOCATIONS:
Overall Officials: JEAN-LUC PERROT, PHD, Principal Investigator — Service de Dermatologie, Hôpital Nord CHU de Saint-Étienne 42055 SAINT-ETIENNE Cedex 2
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Bron
  - Hôpital Nord CHU de Saint-Étienne, Saint-Etienne